CLINICAL TRIAL: NCT06812767
Title: Risk Factors at Chronic Non-communicable Diseases in People of Working Age
Acronym: FORTUNE
Status: Enrolling by invitation | Type: Observational
Sponsor: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Responsible Party: Sponsor
Other Study IDs: 05-05/24
Record Dates: First submitted 2025-02-01; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Chronic Non-communicable Disease
Keywords: arterial hypertension; coronary heart disease; cerebrovascular disease; malignant tumors; chronic obstructive pulmonary disease; asthma; diabetes mellitus; environment; smoking; alcohol consumption; unbalanced diet; hypodynamia; obesity; overweight; dyslipidemia; hyperglycemia; microalbuminuria
MeSH Terms: conditions — Noncommunicable Diseases; Hypertension; Coronary Disease; Cerebrovascular Disorders; Neoplasms; Pulmonary Disease, Chronic Obstructive; Asthma; Diabetes Mellitus; Smoking; Alcohol Drinking; Hypokinesia; Obesity; Overweight; Dyslipidemias; Hyperglycemia | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — blood and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Persons without NCDs: Persons without known NCDs and not using any medication on a permanent basis
  Interventions: Diagnostic Test: electrocardiography; Diagnostic Test: analysis for glucose and cholesterol in the capillary blood; Diagnostic Test: detection of microalbumuria; Diagnostic Test: heart ultrasound examination; Diagnostic Test: carotid artery ultrasound examination

INTERVENTIONS:
Diagnostic Test: electrocardiography — 12 standard leads
Diagnostic Test: analysis for glucose and cholesterol in the capillary blood — express test
Diagnostic Test: detection of microalbumuria — express test
Diagnostic Test: heart ultrasound examination — Ultrasound examination with Lumify Handheld S4-1 Phased Array Ultrasound (Philips)
Diagnostic Test: carotid artery ultrasound examination — Ultrasound examination with Lumify Handheld L12-4 Linear Array Ultrasound (Philips)

SUMMARY:
Objectives: to study the clinical and demographic characteristics of working age persons, to highlight the main factors of non-communicable diseases (NCDs), to identify NCDs with physical examination, laboratory tests, electrocardiography and ultrasound imaging, to develop a corporate prevention program for the company to reduce the risk of complications of NCDs.

Research stages:

1. Questionnaire to identify socio-demographic, behavioral, hereditary, psycho-emotional risk factors of NCDs
2. Laboratory tests (analysis of glucose and cholesterol in the capillary blood, detection of microalbuminuria), diagnostic tests (electrocardiography, and carotid artery ultrasound)
3. Evaluation of the results of questionnaires and surveys. Recommendations for lifestyle modification and follow-up in a local healthcare department

DETAILED DESCRIPTION:
Currently the emphasis in preventive medicine is also on health of the working population, which is a key state policy in the Russian Federation. Health of working citizens is an important factor in the development and safety of the production sector, but it is also the key to health and well-being of all other groups - children and older generations - that is, in fact, the fundamental factor for social development. Therefore, the integration of health-saving technologies into all areas of working life, including production and work activities, is particularly important. In today's world, it is very important that everyone actively participate in the preservation the health of the individual and its high awareness. Awareness of risk factors for chronic non-communicable diseases and measures prevention throughout life is an important part of a healthy society. Monitoring the health of working citizens allows to predict the problem and take the necessary measures in a timely manner.

In the Russian Federation, medical screening is a complex system, including medical examination by physicians of several specialties and application of the necessary methods of examination to identify chronic non-communicable diseases and their risk factors at an early stage that are the main cause of disability and premature mortality in the country's population, and also to form health status groups and provide recommendations for patients. The examination is carried out once every three years and includes a set of methods of advanced examination to identify early on the most likely chronic non-communicable disease for a given age and gender. Regular checkups are the most important mass and highly effective medical technology of health savings.

The work of carrying out regular preventive examinations and check-ups is carried out by primary health care. Often the quality of such work is limited by manpower shortages, technological and logistical barriers. In modern conditions, these obstacles can be overcome by using mobile systems that include modern digital diagnostic technologies, Allow for more in-depth investigation and identification of risk factors not covered by the standard examination protocol. This will increase the coverage and detection of risk factors, which is an important component of the health saving of the working population

ELIGIBILITY:
Inclusion Criteria:

* employees of the company
* persons without NCDs diagnosis and not receiving permanent medication
* residents of the region of the Russian Federation where a factory with permanent or temporary registration is located

Exclusion Criteria:

* refusal to sign informed consent
* any NCDs requiring constant medication
* active cancer
* pulmonary embolism
* valve defects of the heart (except secondary mitral regurgitation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study is planned to include all working citizens who meet the inclusion criteria and have come for preventive examination. In total, at least 2,000 people are planned to be included in the study. All participants will be given informed consent to participate in the clinical trial
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
prevalence of NCDs risk factors | on enrollment
  risk factors of NCDs based on survey results and diagnostic tests
prevalence of NCDs | on enrollment
  diagnosed NCDs based on survey results, and diagnostic tests

SECONDARY OUTCOMES:
Hospitalization | on enrollment
  Urgent or emergent hospitalization during the visit if indicated

CONTACTS AND LOCATIONS:
Overall Officials: Olga Dzhioeva, MD, PhD, Study Director — National Medical Research Center for Therapy and Preventive Medicine
Locations (1):
- National Medical Research Center for Therapy and Preventive Medicine, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided